CLINICAL TRIAL: NCT04869657
Title: Sustainment of Mental Health Supports in Under-Resourced Urban Schools
Brief Title: Sustainment of Mental Health Supports
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: University of Pennsylvania (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 20-018185; 1R01MH122465-01A1 (NIH)
Record Dates: First submitted 2021-04-23; First posted 2021-05-03 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Behavior Disorders
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sustainment 1: Coaches with CHOP Support (Active Comparator): In Year 1 of participation, schools in both arms will receive support for Tier 2 interventions provided by Children's Hospital of Philadelphia (CHOP) research consultants. In Year 2, schools in Sustainment 1 will receive reduced support for Tier 2 interventions provided by school district coaches. The coaches will in turn receive diminished support from research consultants. In Year 3, schools in both conditions will implement Tier 2 interventions with support from school district coaches; coaches will not receive direct assistance from research consultants.
  Interventions: Behavioral: Coaches with Children's Hospital of Philadelphia (CHOP) Research Consultant Support; Behavioral: Coaches without CHOP Research Consultant Support
- Sustainment 2: Coaches without CHOP Support (Active Comparator): In Year 1 of participation, schools in both arms will receive support for Tier 2 interventions provided by CHOP research consultants. In Years 2 and 3, schools in Sustainment 2 will receive support from school district coaches but coaches will not receive help from research consultants.
  Interventions: Behavioral: Coaches without CHOP Research Consultant Support

INTERVENTIONS:
Behavioral: Coaches with Children's Hospital of Philadelphia (CHOP) Research Consultant Support — Coaches employed by the school district will support the implementation of three evidence-based practices, while themselves being remotely supported by CHOP research consultants.
  Arms: Sustainment 1: Coaches with CHOP Support
Behavioral: Coaches without CHOP Research Consultant Support — Coaches employed by the school district will support the implementation of three evidence-based practices without any additional support from CHOP research consultants.

SUMMARY:
Schools are in great need of service delivery systems that can improve school climate and also attend to students' mental health. One effective approach is Positive Behavioral Interventions and Supports (PBIS), a multitiered framework for defining and organizing practices and interventions (including mental health practices).

ELIGIBILITY:
Inclusion Criteria:

* Schools: Any school in the School District of Philadelphia (SDP) already implementing Positive Behavioral Interventions and Supports (PBIS).
* Tier 2 Team Members: Any staff from participating schools involved in the PBIS leadership team at that school.
* Tier 2 Implementers: Any Masters-level staff assigned by their school's principal to deliver Tier 2 interventions.
* Tier 2 Coaches: Any Masters-level clinician employed by the SDP to support staff implementing Tier 2 interventions
* Students: Any student at participating schools in grades 4-8 who scores as eligible for PBIS based on the Social, Academic, and Emotional Behavioral Risk Screener (SAEBRS), which is standard screening criteria in the SDP for Tier 2 services and scores above > 1 SD above the mean on the Emotional Symptoms or Conduct Problems scales of the Strengths and Difficulties Questionnaire (SDQ) plus Impact Supplement scores of 1 (A medium amount) or 2 (A great deal) completed by a parent or a teacher

Exclusion Criteria:

* Schools: Any schools not currently implementing PBIS at Tier 1.
* Tier 2 Team Members and Implementers: Any school personnel that are not involved in the leadership team or tier 2 team.
* Students: Any student with a Special Education classification of "Intellectual Disability;" or with a history of psychotic or autistic spectrum disorders according to school records will be excluded because they would be unlikely to benefit from our tier 2 interventions

Ages: 8 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 392 (Actual)
Dates: Start 2021-09-17 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Fidelity to Tier 2 Interventions Checklists | Up to 14 weeks
  Fidelity will be measured every time a student receives a Tier 2 intervention. All Tier 2 team meetings and child group Tier 2 sessions will be audio-recorded. These recordings will be used to determine content fidelity using the Coping Power, CATS and Check-In/Check-Out Content Fidelity Checklists.
Penetration of Evidence-Based Practices (EBP) | 3 years
  Investigators will assess EBP penetration at the school provider level (behavioral health staff involved in the implementation of EBPs), and at the student service level (students receiving EBPs at Tier 2) during Years 2 and 3 of the study compared to Year 1.This information will be obtained from questionnaires completed by school therapists and their coaches.
Change in the Behavior Assessment System for Children (BASC) from Baseline to Post Intervention | Baseline and 14 weeks (post -intervention)
  Student Mental Health Symptoms will be measured by comparing parental and child scores pre-intervention and post-intervention.The BASC-3 is a 138-item, 4-point, Likert-type rating scale (N=Never, S=Sometimes, O=Often, A=Almost Always) for assessing parental report of child mental health functioning, standardized for ages 2.5 to 18 years.
Change in the Engagement versus Disaffection with Learning from Baseline to Post Intervention. | Baseline and 14 weeks (post-intervention)
  Student Academic Engagement will be measured by comparing teacher and student scores pre-intervention and post-intervention.This is a 20-item, four-point instrument (1 = Not At All True, 2 = Not Very True, 3 = Sort Of True, 4 = Very True) with four sub-scales. Investigators will use the average score for each of the four scales at pre- and post-participation in group cognitive behavioral therapy (CBT) or Check-in/Check-out (CICO).
Cost-effectiveness | up to 5 years
  A Cost Benefit Analysis will be conducted across both sustainment conditions, comparing material expenses, personnel effort, agency and school district salaries, etc. Cost-effective will be measured using qualitative interviews with staff participants.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Eiraldi, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Eiraldi R, McCurdy BL, Khanna MS, Wolk CB, Glick HA, Rabenau-McDonnell QA, Comly R, Rutherford LE, Banks J, Rufe SA, Popkin KM, Wilson T, Henson K, Wandersman A, Jawad AF. Study protocol: cluster randomized trial of consultation strategies for the sustainment of mental health interventions in under-resourced urban schools: rationale, design, and methods. BMC Psychol. 2022 Feb 7;10(1):24. doi: 10.1186/s40359-022-00733-8. PMID 35130964